CLINICAL TRIAL: NCT01543451
Title: Phase II, Double-blind, Randomized, Two-stage, Placebo-controlled Proof of Concept Study in Colorectal Cancer Patients Receiving 5-FU Based Chemotherapy to Assess the Efficacy of Elsiglutide (ZP1846)Administered s.c. in the Prevention of Chemotherapy Induced Diarrhea(CID)
Brief Title: Proof-of-Concept Study in Cancer Patients to Assess Efficacy of Elsiglutide in Preventing Chemotherapy-Induced Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TIDE-11-10
Record Dates: First submitted 2012-02-21; First posted 2012-03-05 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elsiglutide (Experimental)
  Interventions: Drug: Elsiglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elsiglutide — 24 mg administered s.c. once daily for 4 consecutive days from Day 1 chemotherapy
  Arms: Elsiglutide
Drug: Placebo — 24 mg administered s.c. once daily for 4 consecutive days from Day 1 chemotherapy
  Arms: Placebo

SUMMARY:
The main objective of this study will be to obtain data on the efficacy of elsiglutide in preventing Chemotherapy Induced Diarrhea (CID) in patients with colorectal cancer receiving 5-FU based chemotherapy (FOLFOX4 or FOLFIRI regimen) in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Male or female patient ≥ 18 years of age;
3. Confirmed diagnosis of colorectal cancer;
4. Chemotherapy naïve patient;
5. Patient scheduled to receive a FOLFOX4 or FOLFIRI chemotherapy regimen according to the following scheme and dosage (1st cycle):

   AGENT DOSE ROUTE/DURATION DAYS Oxaliplatin or Irinotecan 85/180 mg m2 i.v. infusion/2h 1 FolinicAcid (leucovorin) 200 mg m2 i.v. infusion/2h 1+2 5-Fluorouracil (5FU) 400 mg m2 i.v. bolus 1+2 5-Fluorouracil (5FU) 600 mg m2 i.v. infusion/22h 1+2
6. A performance status of ≤ 2 according to the Eastern Cooperative Oncology Group(ECOG);
7. Non-fertile patient or fertile patient (male or female) using reliable contraceptive measures
8. Female patient of childbearing potential; need to have a negative pregnancy test at screening.

Inclusion criteria 1-8 will be verified at screening.

Inclusion criteria 8 will be re-confirmed on Day 1.

Exclusion Criteria:

1. Inability to understand study procedures and/or cooperate with the study Investigator;
2. Any investigational drugs within 30 days before enrollment in the study or foreseen use of investigational agents during the study;
3. Patient with any type of ostomy;
4. Any previous radiotherapy to the abdomen or pelvis;
5. Scheduled to receive radiotherapy to abdomen or pelvis during the study (Day 1 to Day 14);
6. Scheduled to receive any concomitant chemotherapeutic agent other than FOLFOX4 or FOLFIRI agents (Oxaliplatin, Irinotecan, Folinic acid, 5-FU) from Day 1 to Day 14;
7. Previous use or scheduled to receive monoclonal antibodies (e.g. bevacizumab, cetuximab, etc) during the study (From Day 1 to Day 14);
8. Major surgery within the previous 3 weeks;
9. Any type of condition leading to chronic diarrhea, including but not limited to inflammatory bowel diseases (e.g. ulcerative colitis and Crohn's disease), chronic diarrhea of presumed or confirmed infectious origin and irritable bowel syndrome;
10. Any diarrhea in the 48 hours preceding study drug administration;
11. Use of anti-diarrheal agents within the 48 hours prior to study drug administration;
12. Use of laxatives within 7 days prior to study drug administration;
13. Use of antibiotics within 7 days prior to study drug administration;
14. History of chronic (≥ 30 consecutive days) use of laxatives;
15. Active and ongoing systemic infection;
16. Lactating woman;
17. History of hypersensitivity or allergies to drugs or compounds potentially related to this investigational drug class;
18. Previous exposure to GLP-2 or other compounds in this investigational drug class;
19. Abnormal laboratory values, including

    * Aspartate aminotransferase (AST) ≥ 5 x upper limit of normal
    * Alanine aminotransferase (ALT) ≥ 5 x upper limit of normal
    * Bilirubin > 2 mg/dL (34 μmol/L)
    * Creatinine > 2 mg/dL (177 μmol/L)
    * Albumine < 2 g/dL (20 g/L)
    * Neutrophils< 1.5 x109/L
    * Platelet count < 100 x109/L;
20. Concomitant bleeding disorders;
21. Other serious concomitant illness, which could interfere with the study;
22. Patient who participated in a previous study with elsiglutide (ZP1846).

Exclusion criteria 1-9 and 12-22 will be verified at screening. Exclusion criteria 10 and 11 will be checked on Day 1 only. Exclusion criteria 12, 13 and 15 will be re-checked on Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of Patients experiencing Diarrhea | Day 1 to Day 14
  Severity of Diarrhea will be classified according to the NCI-CTCAE.

SECONDARY OUTCOMES:
Safety and tolerability of the administered repeated doses of elsiglutide (ZP1846) will be evaluated | Day 1 to Day 32
  Safety will be evaluated by monitoring:
  * Physical examination
  * Vital signs
  * Clinical laboratory parameters (hematology, blood chemistry, urinalysis)
  * 12-lead ECG
  * AEs
  * Immunogenicity testing in a subset of patients
PK of elsiglutide will be evaluated | Day 1 to Day 5
  The followin standard PK parameters will be evaluated:
  Tmax, Cmax, AUC0-t, AUC0-24, AUC0-∞, t1/2Z, λZ, CL/F, VZ/F, the effect of multiple dosing will be evaluated (accumulation ratio). Blood sampling for PK will be performed at: pre-dose, 2h, 4, 6, 12, 24 h post-dose

CONTACTS AND LOCATIONS:
Locations (20):
- Bulgaria (4):
  - Department of Chemotherapy, Complex Oncology Center, Rousse, Ruse
  - Chemotherapy Department, Complex Oncology Center, Shumen, Shumen
  - Department of Chemotherapy Specialized Hospital for Active Treatment of Oncological Diseases, Sofia, Sofia
  - Oncology Clinic, Multiprofile Hospital for Active Treatment "Sveta Marina", Varna, Varna
- Hungary (4):
  - Semmelweis University, Department of Diagnostic Radiology and Oncotherapy, Budapest, Budapest
  - Kenezy Hospital, Department of Clinical Pharmacology, Infectology and Allergology, Debrecen, Debrecen
  - Petz Aladar County Teaching Hospital, Center of Oncologic Radiology Hungary, Győr, Hungary
  - Szeged Medical University Department of Oncology and Oncotherapy, Szeged, Szeged
- Romania (5):
  - Fundeni Clinical Institute - Medical Oncology Department, Bucharest, Bucharest
  - Prof. Dr. Ion Chiricuta Institute of Oncology, Medical Oncology Department, Cluj-Napoca, Cluj
  - Euroclinic Oncology Center SRL - Medical Oncology Department, Iași, Iaşi
  - Dr. Constantin Opris Clinical Country Emergency Hospital Baia Mare, Department of Oncology, Baia Mare, Maramureş
  - Sf. Ioan cel Nou Emergency Clincal County Hospital, Suceava, Suceava
- Russia (7):
  - Regional Oncology Center, Arkhangelsk, Arkhangelskaya oblast
  - Kursk Regional Clinical Oncology Center, Kursk, Kursk Oblast
  - Pyatigorsk Oncology Center, Pyatigorsk, Pyatigorsk
  - City #9 Hospital, Saint Petersburg, Sankt-Peterburg
  - City Clinical Oncology Center, Saint Petersburg, Sankt-Peterburg
  - Regional Clinical Oncology Center - Chemotherapy Department, Ulyanovsk, Ulyanovsk Oblast
  - Regional Oncology Hospital, Yaroslavl, Yaroslavl Oblast